CLINICAL TRIAL: NCT03048630
Title: Reducing Chemical Exposures in Nail Salons Using an Owner-to-Worker Intervention
Brief Title: Reducing Chemical Exposures in Nail Salons
Acronym: KHOEDEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cancer Prevention Institute of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2012-008
Record Dates: First submitted 2017-01-31; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Occupational Exposure
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knowledge and behavioral intervention (Experimental): Owner and worker trainings regarding knowledge and behaviors associated with workplace chemical exposure reduction
  Interventions: Behavioral: Education
- Delayed intervention (Other): Delayed knowledge and behavioral intervention
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Owner-to-Worker training about reducing chemical exposures in nail salons

SUMMARY:
In this intervention study, the investigators engage Vietnamese American nail salon owners to train workers within their salons on how to reduce workplace chemical exposures. The long-term goal of the study is to reduce toxic chemical exposures in nail salons and promote worker health and safety in this vulnerable worker population.

DETAILED DESCRIPTION:
The primary hypothesis is that there will be a significantly greater reduction in measured levels of air contaminants among workers in the intervention group than in the comparison group. The primary outcome of interest is workplace chemical exposure reduction.

In addition, the secondary hypotheses are:

1. The proportion of workers who have increased knowledge of workplace chemical exposure reduction (WCER) will be significantly greater in the intervention group than in the comparison group.
2. The proportion of workers who report having modified behavioral and environmental factors that facilitate WCER will increase significantly more in the intervention group than the comparison group.
3. The proportion of workers with decreased work-related health problems will be greater in the intervention group than the comparison group.

As part of the secondary analyses, the investigators will also examine whether changes in knowledge and behavior are associated with workplace chemical exposure reduction and also whether changes in workplace chemical exposure are associated with improved health. The specific aims are to:

1. Enhance existing workplace chemical exposure reduction (WCER) education materials and survey instruments that target Vietnamese nail salon owners and workers.
2. Implement an owner-to-worker intervention to administer the WCER education materials.
3. Evaluate the effectiveness of the owner-to-worker WCER intervention for:

   1. reducing the primary outcome of measured personal levels of air contaminants (e.g., toluene, methyl methacrylate, methyl ethyl ketone, and total volatile organic compounds) in workers;
   2. influencing the secondary outcomes which include:

   i) increasing worker knowledge of WCER

   ii) modifying behavioral and environmental factors that promote WCER

ELIGIBILITY:
Inclusion Criteria:

* Nail salon workers and owners who speak and/or write Vietnamese

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduced measured workplace chemicals by air monitoring | from 4 to 6 months

SECONDARY OUTCOMES:
Behavior and knowledge change by questionnaire | from 4 to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Prevention Institute of California, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No